CLINICAL TRIAL: NCT01682785
Title: Incidence and Prevalence of and Factors Associated With Metabolic Syndrome and Thyroid Dysfunction in Patients With Major Depressive Disorder
Brief Title: Incidence of Metabolic Syndrome and Thyroid Dysfunction in Patients With Major Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Chawanun Charnsil, Asso. prof., Chiang Mai University
Other Study IDs: MDD-Met
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Major Depressive Disorder; Metabolic Syndrome; Thyroid Dysfunction
Keywords: Major depressive disorder; Metabolic syndrome; Thyroid dysfunction; incidence
MeSH Terms: conditions — Depressive Disorder, Major; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Aim 1 is to study prevalence and 1 year incidence of metabolic syndrome in major depressive disorder and factors correlation.

Aim 2 is to study prevalence and 1 year incidence of thyroid dysfunction in major depressive disorder and factors correlation.

ELIGIBILITY:
Inclusion Criteria:

* patient with major depressive disorder
* age over 18 years

Exclusion Criteria:

* subject who cannot give information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major depressive disorder
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2012-09